CLINICAL TRIAL: NCT01186679
Title: Surgical Transplantation of Autologous Bone Marrow Stem Cells With Glial Scar Resection for Patients of Chronic Spinal Cord Injury and Intra-thecal Injection for Acute and Subacute Injury - A Preliminary Study
Brief Title: Safety and Efficacy of Autologous Bone Marrow Stem Cells in Treating Spinal Cord Injury
Acronym: ABMST-SCI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Stemcell Services Limited (Industry)
Responsible Party: Dr.SGA.Rao, Chairman, International Stemcell Services Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSL-AuBM-SCI
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Laminectomy; Injections, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intralesional (Experimental): 1. Surgical transplantation into the lesion site in chronic patients
  2. Direct intrathecal implantation in acute and subacute patients
  Interventions: Procedure: laminectomy
- intrathecal (Experimental): direct into the CSF through lumbar puncture
  Interventions: Procedure: Intrathecal

INTERVENTIONS:
Procedure: laminectomy — surgical laminectomy with glial scar resection
  Arms: Intralesional
Procedure: Intrathecal — direct into the CSF through lumbar puncture
  Arms: intrathecal

SUMMARY:
The projected data related to the burden of spinal cord injuries induced limb paralysis in India is quite alarming. This is attributed to the rapid industrialization and economical development in the country. Increase in vehicular traffic has caused numerous road traffic accidents. Rapid increase in populations, development in the computer technology and real estate business lead to construction of huge buildings which indirectly adds to the injuries due to fall. Spinal cord injuries could not be treated adequately with the prevailing treatment modalities. In view of this, there is definitely an urgent need for finding different methods of treatment for these patients who cannot undergo established modalities of treatment or these have been tried unsuccessfully. Since a large number of these patients will loose their productive life and at the prime of their lives, one such alternate therapy, which seems to offer some promise, is "stem cell" therapy, which has been well studied and published in prestigious journals.

In our present study, we want to evaluate the safety and efficacy of autologous bone marrow derived stem cells surgically transplanted directly into the lesion site with glial scar resection for 8 indian patients of chronic spinal cord injury and intra-thecal injection for 4 indian patients of acute and subacute injury.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to give voluntary (patients may not be able to write) consent.
2. Must be able to understand study information provided to him.
3. Patients with complete spinal cord trans-section: at least post 6 months after spinal cord Injury (in chronic patients), < 2 weeks in acute category and 2-8 weeks in subacute patients.
4. The level of spinal cord injury must be between C4 and T12(neurological level)
5. Spinal cord injury categorized in terms of ASIA Impairment scale.
6. Age should be between 20-55 years

Exclusion Criteria:

* Mechanical ventilation due to neurological impairment
* Multiple level trauma
* Undetermined size and location of Spinal Cord injury
* Gunshot or other penetrating trauma to the spinal cord
* Longitudinal dimension of injury by MRI is greater than 3spinal segments
* Associated severe head injury
* More than 9cms long bone fracture
* Women who are pregnant or lactating
* Serious pre-existing medical conditions
* Disease or impairment that precludes adequate neurological examination.
* Should not have co-morbidities like Diabetes, Systemic Hypertension etc.
* Severe co-morbidities/bed sores Tests positive for infectious diseases Deranged Coagulation profile and Hb < 8mg/dl

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with adverse events as a measure of safety and tolerability. Significant clinical improvement in ASIA impairment scale and general condition | 18 months
  American Spinal Injury Assessment scale of A,B,C,D or E

SECONDARY OUTCOMES:
Changes in the MRI, Neurological improvement (cranial/spinal reflexes) and evoked potentials study | 18 months
  MRI findings of the lesion, Nerve conduction studies of the region and somatosensory evoked potentials of the same region

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Arvind Bhateja, MCh.Neurosurgery, Principal Investigator — Sita Bhateja Speciality Hospital
Locations (1):
- Sita Bhateja Speciality Hospital, Bangalore, Karnataka, India